CLINICAL TRIAL: NCT03356418
Title: Immediate Effects of Whole-Body Vibration on Neuromuscular Performance and Postural Control in Elderly: A Randomized Controlled Trial
Brief Title: Immediate Effects of Whole-Body Vibration on Neuromuscular Performance and Postural Control in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Jamilson Simões Brasileiro, Associeted Professor and Researcher, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DL2017.2
Record Dates: First submitted 2017-11-19; First posted 2017-11-29 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Neuromuscular Performance and Balance
Keywords: Exercise; Vibration; Torque; Aging
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WBV exercise group (Experimental): Subjects will perform an isometric semi-squat exercise associated with the vibratory platform. The exercise will consist of 4 series of an isometric half-squat exercise with 1 minute and a half of duration and a rest interval of 1 minute. The vibratory platform will be connected at the beginning of each series, set at a vibration frequency of 40 Hertz (Hz) and peak-to-peak amplitude of 4 millimeters (mm) resulting in a peak acceleration of 128 ms2 (12.8 g). This should provide the equivalent of 3600 vertical vibrations, totaling 14400 vibrations per training session
  Interventions: Other: WBV exercise group
- Sham WBV exercise group (Sham Comparator): Subjects will perform an isometric semi-squat exercise associated with the vibratory platform. The exercise will consist of 4 series of an isometric half-squat exercise with 1 minute and a half of duration and a rest interval of 1 minute. The vibratory platform will remain off at all sessions. A device will be attached to the side of the platform in order to produce a sound, similar to the sound produced by the vibrating platform when it is in operation.
  Interventions: Other: Sham WBV exercise group

INTERVENTIONS:
Other: WBV exercise group — The intervention will consist of a half-squat isometric whole-body vibration exercise with the platform configured at a frequency of 40 Hz and peak-to-peak amplitude of 4 mm. The sessions will be held 2 times a week, consisting of 4 sets of 1 and a half minutes of exercise on the platform. Rest intervals of 1 minute between sets will be respected.
  Arms: WBV exercise group
Other: Sham WBV exercise group — The intervention will consist of as half-squat isometric exercise , but the platform will remain off at all sessions. A device will be attached to the side of the platform in order to produce a sound, similar to the sound produced by the vibrating platform when it is in operation.
  Arms: Sham WBV exercise group

SUMMARY:
The purpose of this study is to analyze the immediate effects of an exercise protocol on the vibration platform on the functional and neuromuscular performance of lower limbs, postural control and life quality in healthy elderly.

DETAILED DESCRIPTION:
The research is a randomized controlled trial that will be developed at the Laboratório de Análise da Performance Muscular (LAPERN) of the Physiotherapy Department of the Federal University of Rio Grande do Norte (UFRN). The population of the present study will be formed by elderly individuals living in the city of Natal / RN, aged between 65 and 75 years, of both sexes, without distinction of race, education and marital status. The research sample will be of a non-probabilistic type, in which these will be allocated randomly into two distinct groups: placebo group (GP) and experimental group (GE). This research was submitted to the Research Ethics Committee (CEP) for UFRN through the national interface Plataforma Brasil. The present research contemplates the ethical aspects based on Resolution 466/2012 of the National Health Council (CNS) and the Declaration of Helsinki for research with humans. In addition, the survey will be recorded in Clinicals Trial. All data will be recorded in a database of the laboratory under confidentiality and can only be handled by the responsible researchers. The study will only begin after the issuance of the referent opinion approving the project. All subjects will be duly informed and instructed regarding the scheduled procedures, which will only be executed after reading, accepting and signing the Term of Free and Informed Consent (TFIC). After approval by the Research Ethics Committee, following resolution 466/2012, a pilot study was carried out aiming at the adequacy of all the research procedures, as well as the training of the researchers involved. Initially the research will begin with the selection of the sample according to the inclusion criteria descried elsewhere. The evaluation will be scheduled by telephone contact. Following this, the volunteers will receive the TFIC for reading and due signature. The data collection process will take place in four stages: (1) initial evaluation, (2) sample allocation (3) application of exercise program and (4)reevaluation. The evaluations will be composed by the dynamometric analysis associated with EMG (electromyography) and postural control analysis. The volunteers will be allocated randomly into 2 groups: placebo group (with the platform off) or experimental group (with the platform set at a frequency of 40 Hz and amplitude of 4 mm). Both will perform a bout of exercise in the vibrating platform, consisting of a static bipodal squat at 40 ° of knee flexion, with 4 sets of 1.5 min, with a rest interval of 1 minute. Immediately after the exercise the volunteers will be submitted to a revaluation, with the same procedures of the initial evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Both genders;
* Exhibiting ankle, hip and knee joint integrity of the non-dominant limb;
* No history of muscle or joint injuries in the assessed limb in the last 6 months, or neurological, visual and/or non-corrected auditory impairments;
* Do not have metallic implants in the lower limbs;
* Do not have decompensated and / or untreated cardiovascular diseases;
* Do not have advanced osteoporosis;
* Do not have neurodegenerative diseases;
* Do not have vestibular disorders;
* Do not have uncorrected visual or hearing deficits.

Exclusion Criteria:

* Elderly classified as very active or active;
* Report cardiac and / or respiratory discomfort, nausea, vertigo and pain during during the evaluations and exercise sessions;
* Do not understand and do not correctly perform the commands offered in the assessment and / or intervention protocols;

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Change in average power measured through isokinetic dynamometer | Baseline and immediately after the intervention protocol.
  Measured through isokinetic dynamometry. The analyzed variable will be average power (in watts).

SECONDARY OUTCOMES:
Change in Muscle activation measured through surface electromyography | Baseline and immediately after the intervention protocol.
  Measured by surface electromyography. The analyzed variable will be the amplitude of muscle activation (in microvolts).
Change in Balance measured through baropodometry | Baseline and immediately after the intervention protocol .
  Measured by baropodometry. The analyzed variable will be the oscilation of center of pressure (in mm).
Change in peak torque normalized by body weight measured through isokinetic dynamometer | Baseline and immediately after the intervention protocol.
  Measured through isokinetic dynamometry. The analyzed variable will be a combination of peak torque normalized by body weight (in percentage).
Change in total work measured through isokinetic dynamometer | Baseline and immediately after the intervention protocol.
  Measured through isokinetic dynamometry. The analyzed variable will be total work (in joules).
Change in peak torque measured through isokinetic dynamometer | Baseline and immediately after the intervention protocol.
  Measured through isokinetic dynamometry. The analyzed variable will be peak torque (in Newtons).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Borges, MS, Principal Investigator — Universidade Federal do Rio Grande do Norte; Lidiane C Bulhões, Esp, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal University of Rio Grande do Norte (UFRN), Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No